CLINICAL TRIAL: NCT04501471
Title: The Rural African American's Health Project
Acronym: RAAFHP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Gene H. Brody, Regents Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2006-10685
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: SAAF-T; FUEL for Families

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and providers were not aware that the Fuel condition was considered an attention control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAAF-T (Experimental): Participants received a 5 session, 10-hour family centered prevention program designed to prevent substance use, conduct problems, and risky sexual behavior
  Interventions: Behavioral: SAAF-T
- Fuel for Families (Placebo Comparator): Participants received a 5 session, 10 hour family centered program that focused on healthy nutrition and exercise.
  Interventions: Behavioral: Fuel for Families

INTERVENTIONS:
Behavioral: SAAF-T — Parents and youth meet separately during first hour to engage in activities then meet in family groups during the second hours of each session.
  Other Names: Strong AFrican American Families-Teen Program
  Arms: SAAF-T
Behavioral: Fuel for Families — Parents and youth meet separately during first hour to engage in activities then meet in family groups during the second hours of each session.
  Arms: Fuel for Families

SUMMARY:
This is an attention controlled randomized clinical trial testing the efficacy of the Strong African American Families-Teen program. The two arm trial tests SAAF-T, a family centered brief intervention against a similarly designed program that targets nutrition and exercise. The outcomes examined include substance use and risky sexual behavior.

DETAILED DESCRIPTION:
In the past, African American adolescents in rural areas have avoided the high-risk behaviors prevalent among youth in urban areas. Recent epidemiologic data, however, indicate that rural African American youth use substances and engage in high-risk sexual behavior at rates equal to or exceeding those in densely populated inner cities (Kogan, Berkel, Chen, Brody, & Murry, in press; Milhausen et al., 2003). These risk behaviors predict HIV infection, adolescent parenthood, school dropout, involvement with the criminal justice system, and continued substance use during early adulthood (Friedman et al., 1996; Miller, Boyer, & Cotton, 2004; St. Lawrence & Scott, 1996; Tucker, Orlando, & Ellickson, 2003). No developmentally appropriate, culturally sensitive prevention programs have been developed to deter substance use and high-risk sexual behavior among the several million African American adolescents who live in the rural South (Murry & Brody, 2004). To address this public health need, Drs. Brody and Murry from the University of Georgia and Drs. DiClemente and Wingood from Emory University designed a multicomponent, family-centered prevention program, the Strong African American Families-Teen program (SAAF-T). We conducted a randomized prevention trial to test the program's efficacy. The sample included 502 rural African American families with a 10th-grade student, half of whom will be assigned randomly to a prevention group and half to an attention-control group. Pre-intervention, post-intervention, and long-term follow-up assessments of adolescents' substance use and high-risk sexual behavior were gathered from the entire sample. Specific aims were to test hypotheses that rural African American adolescents randomly assigned to participate in SAAF-T, compared to attention-control participants, will demonstrate lower rates of substance use and risky sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Black or African American
* 10th grade in public school in targeted county

Exclusion Criteria:

* Unable to participate in group-based intervention due to mental health

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 502 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Substance Use | Follow up period baseline to 22 months post-baseline
  Index of alcohol, cigarette, and marijuana use in the past 3 months
Risky Sexual Behavior | Follow up period baseline to 22 months post-baseline
  Count of unprotected intercourse

SECONDARY OUTCOMES:
Depressive symptomology- CES-D Scale | Symptoms in past week assessed, follow up period includes baseline to 22 months post baseline
  Symptoms of depression, 20 items
Conduct Problems | Follow up period baseline to 22 months post-baseline
  Using 14 questions from the National Youth Survey,adolescents indicated the frequency during the past 6 months with which they had fought, stolen, been truant from school, or been suspended from school. Adolescents' responses were summed, and the sum constituted the conduct problems score.13

OTHER OUTCOMES:
Discussion Quality Scale | Follow up period -baseline to 6 month posttest
  The DQS assessed communication frequency and quality for discussions of difficult issues.
Family Support Inventory | Follow up period -baseline to 6 month posttest
  The FSI measured provision of emotional support, involvement, and quality of caregiver-youth communication

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data

REFERENCES:
- [Derived] Brody GH, Yu T, Chen E, Miller GE, Barton AW, Kogan SM. Family-Centered Prevention Effects on the Association Between Racial Discrimination and Mental Health in Black Adolescents: Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2021 Mar 1;4(3):e211964. doi: 10.1001/jamanetworkopen.2021.1964. PMID 33760092